CLINICAL TRIAL: NCT05721872
Title: An Exploratory Phase I/II Single-center Clinical Trial of the Efficacy, Tolerability and Safety of Intravenous D-isoascorbic Acid With Arsenic Trioxide in Patients With Advanced/Metastatic Colorectal Cancer Who Have Exhausted Standard Therapy
Brief Title: Efficacy, Tolerability and Safety of Intravenous D-VC With ATO in Patients With Advanced/Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nazarbayev University (Other)
Collaborators: National Laboratory Astana (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR11765589
Record Dates: First submitted 2023-01-18; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Colorectal Cancer; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combination of D-isoascorbic acid (D-VC) with arsenic trioxide (ATO)-Phase 1 (Experimental): Participants will receive single intravenous administration as monotherapy of D-isoascorbic acid (D-VC) with dose escalation (0.05, 0.1, 0.2 g/kg/day) and with arsenic trioxide (ATO).
  Patients who have satisfactorily tolerated the study drug in combination with arsenic trioxide (ATO) in a phase I study are transferred to a phase II clinical trial.
  Interventions: Combination Product: D-isoascorbic Acid (D-VC) With Arsenic Trioxide (ATO)
- Combination of D-isoascorbic acid (D-VC) with arsenic trioxide (ATO)-Phase 2 (Experimental): After 2 hours of intravenous administration of arsenic trioxide (ATO) (at a dose of 0.15 mg / kg / day) participants will further receive D-isoascorbic acid (D-VC) intravenously once a day at the maximum tolerated dose, determined at the end of phase I.
  Interventions: Combination Product: D-isoascorbic Acid (D-VC) With Arsenic Trioxide (ATO)
- Standard therapy (FOLFOX/FOLFIRI)-Phase 2 (Active Comparator): Drug: FOLFOX/FOLFIRI regimen FOLFOX - oxaliplatin 85mg/m2 1 day, Leucovorin 200mg/m2 IV 2h, 1, 2 days, 5 - Fluorouracil 400mg/m2 IV bolus, 1, 2 days, 5 - Fluorouracil 600mg/m2 IV 22h, 1, 2 days
  FOLFIRI - Irinotecan 180 mg/m2 IV, Leucovorin 400 mg/m2 IV, Fluorouracil bolus 400 mg/m2 IV, Fluorouracil infusional 2400 mg/m2 IV. Courses are held every 2 weeks
  Interventions: Drug: FOLFOX/FOLFIRI regimen

INTERVENTIONS:
Combination Product: D-isoascorbic Acid (D-VC) With Arsenic Trioxide (ATO) — After 2 hours of intravenous administration of arsenic trioxide (ATO) (at a dose of 0.15 mg / kg / day) participants will further receive D-isoascorbic acid (D-VC) intravenously once a day at the maximum tolerated dose, determined at the end of phase I.
  Phase 1 - Scheme 1 - single intravenous administration in monotherapy with dose escalation (0.05, 0.1, 0.15 g/kg/day); Scheme 2 - single intravenous administration in the mode of sequential administration with arsenic trioxide with dose escalation of D-isoascorbic acid (0.05, 0.1, 0.15 g/kg/day).
  Phase 2 - Study group 1: After 2 hours of intravenous administration of arsenic trioxide (ATO) (at a dose of 0.15 mg / kg / day) participants will further receive D-isoascorbic acid (D-VC) intravenously once a day at the maximum tolerated dose, determined at the end of phase I for at least 15 patients.
  Arms: Combination of D-isoascorbic acid (D-VC) with arsenic trioxide (ATO)-Phase 1; Combination of D-isoascorbic acid (D-VC) with arsenic trioxide (ATO)-Phase 2
Drug: FOLFOX/FOLFIRI regimen — FOLFOX - oxaliplatin 85mg/m2 1 day Leucovorin 200mg/m2 IV 2h, 1, 2 days 5 - Fluorouracil 400mg/m2 IV bolus, 1, 2 days 5 - Fluorouracil 600mg/m2 IV 22h, 1, 2 days
  FOLFIRI Irinotecan 180 mg/m2 IV Leucovorin 400 mg/m2 IV Fluorouracil bolus 400 mg/m2 IV Fluorouracil infusional 2400 mg/m2 IV Courses are held every 2 weeks
  Arms: Standard therapy (FOLFOX/FOLFIRI)-Phase 2

SUMMARY:
The goal of this exploratory phase I/II single-center clinical trial is to evaluate effectiveness, tolerability, and safety of Intravenous D-isoascorbic Acid (D-VC) With Arsenic Trioxide in Patients With Advanced/Metastatic Colorectal Cancer Who Have Exhausted Standard Therapy The main questions are to learn about effectiveness, tolerability, and safety of Intravenous D-isoascorbic Acid (D-VC) With Arsenic Trioxide.

The study aims to:

1. Assess the tolerability and pharmacokinetics of D-isoascorbic acid (D-VC) with a single intravenous injection in the monotherapy regimen and in the sequential administration regimen with arsenic trioxide (ATO) in patients on standard therapy for advanced/metastatic malignancies (Phase I)
2. Evaluate the efficacy and safety of D-isoascorbic acid (D-VC) with repeated intravenous administration in the mode of sequential administration with arsenic trioxide (ATO) in patients who have exhausted standard therapy for advanced/metastatic colorectal cancer (Phase II)

In phase I participants will receive single intravenous administration as monotherapy of D-isoascorbic acid (D-VC) with dose escalation (0.05, 0.1, 0.2 g/kg/day) and with arsenic trioxide (ATO).

Patients who have satisfactorily tolerated the study drug in combination with arsenic trioxide (ATO) in a phase I study are transferred to a phase II clinical trial.

To study the safety and efficacy of the study drug in phase II, D-VC after the administration of ATO will be implemented in 2 groups:

Study group 1: ATO (at a dose of 0.15 mg / kg / day) after intravenous administration after 2 hours D-VC intravenously once a day at the maximum tolerated dose, determined at the end of phase I for at least 15 patients.

Group 2 standard therapy: 15 patients.

For the phase I researchers will compare laboratory tests (including clinical biochemistry and hematology), vital signs, clinical adverse events (diseases, symptoms and complaints) and other specific safety tests (for example, an electrocardiogram, ophthalmic examination) between groups. They will also measure the degree to which overt adverse reactions can be subjectively tolerated by the subject of the study.

For the phase II researchers will compare degrees of tumor volume reduction on CT; objective response rate (ORR) based on BICR according to RECIST v1.1 between test and standard therapy groups. They will also continue evaluation of safety and tolerability of ATO + D-VC combination therapy.

ELIGIBILITY:
Phase 1:

INCLUSION CRITERIA:

* informed consent to participate in the study
* patients of the second clinical group with malignant neoplasms of a common/metastatic form that have exhausted standard therapy.
* patients who have received at least 3 lines of standard therapy, including those with the use of targeted drugs, patients who have exhausted the possibilities of using specialized drugs, as part of the recommendations of treatment protocols
* the presence of "+" KRAS / NRAS status of the primary tumor or metastatic focus (determined in LEKzone 2, codons 12, 13, 61)
* ≥1 measurable lesion defined by RECIST v1.1
* ECOG PS 0.1 or 2

EXCLUSION CRITERIA:

* age up to 18 years
* pregnancy and lactation
* patients with an autoimmune disease or with a medical diagnosis requiring systemic immunosuppression
* decompensated diabetes mellitus
* renal failure, urolithiasis
* diabetes
* thrombophlebitis, tendency to thrombosis
* severe lung disease, dyspnea at rest, pleural effusion
* cardiovascular insufficiency, ejection fraction of the heart <40%
* sensory neuropathy of the 1st degree of any etiology
* uncontrolled infections
* persons from the category of "vulnerable patients" (homeless, military personnel, incapacitated, patients in emergency conditions, other persons who may be subjected to pressure);
* Allergy in history and during screening (drug, pollen, etc.);
* participation in any other clinical trial;
* hypersensitivity to arsenic;
* individual intolerance to ascorbic acid;
* thrombophlebitis and thrombosis, a tendency to thrombosis in history;
* increased blood clotting and pathologies associated with this deviation;
* diabetes;
* nephrolithiasis or nephrolithiasis;
* the patient does not agree to perform the procedures required by the protocol and is unable to adhere to the schedule of procedures.
* if the patients have any other laboratory or other abnormalities, in the opinion of the Investigator, that can harm the patients and the results of the study.

Phase II:

INCLUSION CRITERIA:

for both groups (30 patients, considering 20% decrease from the study):

* informed consent to participate in the study
* patients of the second clinical group with advanced/metastatic colorectal cancer
* Patients must have previously received at least 3 lines of standard drug therapy, including those with the use of targeted drugs, who have exhausted the possibilities of using specialized drugs, as part of the recommendations of colorectal cancer treatment protocols - the presence of "+" KRAS / NRAS status of the primary tumor, or metastatic focus (determined in exon 2, codons 12, 13, 61)
* ≥1 measurable lesion defined by RECIST v1.1
* ECOG PS 0.1 or 2

EXCLUSION CRITERIA:

* age up to 18 years
* patients with an autoimmune disease or with a medical diagnosis requiring systemic immunosuppression
* decompensated diabetes mellitus
* renal failure, urolithiasis
* thrombophlebitis, tendency to thrombosis
* severe lung disease, dyspnea at rest, pleural effusion
* cardiovascular insufficiency, ejection fraction of the heart <40%
* sensory neuropathy of the 1st degree of any etiology
* uncontrolled infections
* persons from the category of "vulnerable patients" (homeless, military personnel, incapacitated, patients in emergency conditions, other persons who may be subjected to pressure);
* Allergy in history and during screening (drug, pollen, etc.);
* participation in any other clinical trial;
* hypersensitivity to arsenic;
* individual intolerance to ascorbic acid;
* thrombophlebitis and thrombosis, a tendency to thrombosis in history;
* increased blood clotting and pathologies associated with this deviation;
* diabetes;
* nephrolithiasis or nephrolithiasis;
* the patient does not agree to perform the procedures required by the protocol and is unable to adhere to the schedule of procedures.
* if the patients have any other laboratory or other abnormalities, in the opinion of the Investigator, that can harm the patients and the results of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline DV-C levels at 1 hour | Baseline, 1 hour
  Patients who have satisfactorily tolerated D-isoascorbic Acid (D-VC) in combination with arsenic trioxide (ATO) in a phase I study are transferred to a phase II clinical trial.
Change from baseline DV-C levels at 3 hours | Baseline, 3 hours
  Patients who have satisfactorily tolerated D-isoascorbic Acid (D-VC) in combination with arsenic trioxide (ATO) in a phase I study are transferred to a phase II clinical trial.
Change from baseline DV-C levels at 6 hours | Baseline, 6 hours
  Patients who have satisfactorily tolerated D-isoascorbic Acid (D-VC) in combination with arsenic trioxide (ATO) in a phase I study are transferred to a phase II clinical trial.
Change from baseline DV-C levels at 24 hours | Baseline, 24 hours
  Patients who have satisfactorily tolerated D-isoascorbic Acid (D-VC) in combination with arsenic trioxide (ATO) in a phase I study are transferred to a phase II clinical trial.
Response to D-isoascorbic Acid (D-VC) in combination with arsenic trioxide (ATO) | Baseline, 4 weeks
  Objective partial or complete response by RECIST 1.1, confirmed on a second CT scan at least 4 weeks apart

SECONDARY OUTCOMES:
Change from baseline number of participants with treatment-related adverse events as assessed by CTCAE v4.0 at 1 hour | Baseline, 1 hour
  Adverse events in patients will be assessed by CTCAE v4.0
Change from baseline number of participants with treatment-related adverse events as assessed by CTCAE v4.0 at 3 hours | Baseline, 3 hours
  Adverse events in patients will be assessed by CTCAE v4.0
Change from baseline number of participants with treatment-related adverse events as assessed by CTCAE v4.0 at 6 hours | Baseline, 6 hours
  Adverse events in patients will be assessed by CTCAE v4.0
Change from baseline number of participants with treatment-related adverse events as assessed by CTCAE v4.0 at 24 hours | Baseline, 24 hours
  Adverse events in patients will be assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Kazakh Institute of Oncology and Radiology, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: No